CLINICAL TRIAL: NCT05118971
Title: Comparison of Muscle Activity in Exercise Bike and Elliptical Trainer in Individuals With Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Collaborators: Douglas Haselstrom (Unknown)
Responsible Party: Principal Investigator, Fernanda Cechetti, Doutora, Federal University of Health Science of Porto Alegre
Other Study IDs: FUHSPortoAlegrePriscila
Record Dates: First submitted 2021-05-10; First posted 2021-11-12 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injuries; Motor Activity; Electromyography; Physical Therapy
MeSH Terms: conditions — Spinal Cord Injuries; Motor Activity

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- elliptical (GE): The patient is suspended supported by the hip positioner, secured by nylon straps to a galvanic iron grid fixed to the ceiling with parabolts. The height of the seat belts will be measured according to the patient's proper position in the device. The weight support belt will be adjusted to maximize load bilaterally without knee deformation during correct posture, manual assistance will be provided by physical therapists on each leg. A physical therapist's hand will be placed on the anterior surface of the leg below the patella to aid in knee extension during the elliptical gait simulation. The other hand will be placed on the ankle to aid in the movement of the feet during the alternating movement of the legs and the return of the heel placement to the starting position. The patient performs the movements at the maximum speed he can, recording the electromyographic signal of the selected muscles for 20 seconds.
  Interventions: Diagnostic Test: muscle activation of the vastus lateralis, vastus medialis, gluteus medius, tibialis anterior, rectus abdominis and paravertebral muscles
- elliptical with biofeedback (GEB): The same described in the elliptical group adding biofeedback.
  Interventions: Diagnostic Test: muscle activation of the vastus lateralis, vastus medialis, gluteus medius, tibialis anterior, rectus abdominis and paravertebral muscles
- bicycle (GB): The patient will have the help of two physiotherapists to position themselves, who will also assist in pedaling as needed. The patient will also be asked to perform the movements at the maximum speed he can, recording the electromyographic signal of the same selected muscles for 20 seconds.
  Interventions: Diagnostic Test: muscle activation of the vastus lateralis, vastus medialis, gluteus medius, tibialis anterior, rectus abdominis and paravertebral muscles
- bike with biofeedback (GBB): The patient will have the help of two physiotherapists to position themselves, who will also assist in pedaling as needed. The patient will also be asked to perform the movements at the maximum speed he can, recording the electromyographic signal from the same selected muscles for 20 seconds, adding biofeedback.
  Interventions: Diagnostic Test: muscle activation of the vastus lateralis, vastus medialis, gluteus medius, tibialis anterior, rectus abdominis and paravertebral muscles

INTERVENTIONS:
Diagnostic Test: muscle activation of the vastus lateralis, vastus medialis, gluteus medius, tibialis anterior, rectus abdominis and paravertebral muscles — understand the pattern of muscle activation during modalities used in this study with the selected population, it becomes extremely important, allowing the quantification of muscle functions and, therefore, prescribing exercises more adequately to achieve therapeutic goals.

SUMMARY:
Spinal cord injury is caused by any harmful process in the spinal cord, impairing its function, generating loss of muscle strength, impairing orthostatism and walking. In rehabilitation, some strategies are used to activate the muscles involved in the gait of these individuals, including the ergometric bicycle and the elliptical. Understanding the pattern of muscle activation generated by these methods is important to answer questions arising from clinical practice. Thus, we seek to verify the pattern of muscle activation of the vastus laterals, vastus medialis, gluteus medius, tibialis previous, rectus abdominis and paravertebral muscles during exercises with ellipticals and ergometric bicycle with and without electromyography biofeedback in individuals with spinal cord injury. Cross-sectional study of the type crossover. Individuals will sign the Informed Consent Form (FICF) and answer the identification form. They will be evaluated for functionality using the Functional Independence Measure (FIM), injury classification by the American Spinal Injury Association (ASIA) and muscle tone by the modified Ashworth scale. Later, they will be randomized to define the order of the devices in which they will be evaluated. Muscle activity will be verified with electromyography of the paravertebral, abdominal, vastus laterals, vastus medialis, gluteus medius and tibialis anterior unilateral muscles on the right side of individuals, comparing muscle activation during exercise cycling, elliptical and adding biofeedback in both modalities. The wash-out interval between each evaluation will be 7 days. We hypothesize that the elliptical with biofeedback will cause greater activation of the assessed muscles.

DETAILED DESCRIPTION:
Spinal cord injury is caused by any mechanism of injury that attacks and impairs the integrity of the spinal cord, preventing it from performing its functions.

It is estimated that the incidence of spinal cord trauma in Brazil is greater than 10,000 new cases per year, 80% being men and 60% aged between 10 and 30 years, with trauma being the predominant cause.

Initial trauma causes injuries by mechanical force, which can cause damage by compression, laceration or section. Any damage to this structure triggers an inflammatory response with edema and, consequently, ischemia, gradually aggravating the injury process, compromising neuronal homeostasis.

The ASIA scale is globally standardized to assess the type of injury. With this scale it is possible to assess the sensory levels preserved through the corresponding dermatomes at each level, testing the superficial and deep sensitivity below the level of the lesion. Motor level is assessed by myotomes, grading the strength of each muscle corresponding to spinal levels.

Neurological disorders resulting from spinal cord injury compromise motor, sensory and autonomic functions, resulting in total or partial loss of voluntary muscle activity, sensitivity, functioning of the urinary, intestinal, respiratory, circulatory and reproductive systems. At the corresponding level, epicritic sensitivity is preserved as it courses in the ipsilateral posterior funiculus. There will also be loss of painful and thermal sensations due to disruption of the nerve fibers that cross the white commissure.

Muscle weakness is the most limiting impairment caused by neurological damage. There is a limitation of activity and several restrictions, which influence the quality of life. The deficit in muscle strength leads to limitations in performing a series of functional activities. The strength of major muscles or muscle groups contributes to functional capacity. Functional independence is positively associated with the peak torque performed by the muscles used to perform a given task.

Physiotherapy has an essential role in the acute and chronic care of these patients, acting as a guide, promoting a greater level of independence, and should aim at preventing deformities, modulating muscle tone, enhancing respiratory muscle function, using various techniques such as transfer training, postural changes, wheelchair handling, balance training, orthostatism and, within the patient's functional potential, restoration of gait and lower limb function, benefiting the performance of activities of daily living, and quality of life.

In spinal cord injury, the deficit of muscle activation compromises many functional actions such as the development of gait, but there are encouraging results with physical therapy techniques that are effective in improving the prognosis of locomotor movement.

Therefore, a set of factors influence gait, which results from an interaction and organization of the neural and mechanical systems, in addition to musculoskeletal dynamics, modulation of the upper nervous system and the afferent pathway, which is also controlled by the Central Pattern Generator through a programming based on a predetermined spinal circuit, capable of producing a rhythm associated with gait.

The Central Pattern Generator is a network of neurons that can produce a variety of movement activity, responsible for automating gait, which depends on feedback from proprioceptors and higher nerve interactions. This generator is responsible for rhythmic motor patterns, generated by inhibitory and excitatory processes of the lower limbs during movements. There is an excitatory and inhibitory relay between agonist and antagonist muscles alternating between limbs.

In these patients, this neuronal domain is compromised, making it difficult to modulate muscle activation. However, recent studies have suggested the existence of effective responses in locomotor training with partial body weight support, leading to an improvement in locomotor patterns.

Locomotor training with partial weight bearing for neurological patients has been studied and considered an important therapeutic mechanism in order to reduce the effects caused by changes in spinal cord injury, being able to fully explore the activation of the patient's potential inducing neural plasticity, providing motor related relearning to the specific task.

Locomotor exercises are based on standardized neural activity. Process by which the central nervous system develops its structure and function in human growth. Continuous repetition of movement can help create this neural pattern in the brain and spinal cord.

There are some devices used in the physiotherapy routine that work rhythmically, for locomotor training and activation of several muscles recruited in the performance of these motor tasks, including the elliptical and the bicycle.

The elliptical is a walking simulator and can also be used for this purpose, which is advantageous in this modality as it reduces the impact on joints, benefiting individuals with impaired balance, as the feet remain in continuous contact with the support surface.

The elliptical provides training with cyclic movement, alternating the lower limbs through a system of levers and sliding axles. When compared to walking on a treadmill, studies suggest that the elliptical reduces plantar pressure in the contact phase of the heel, in addition to reducing the impact of the foot with the contact surface, increasing muscle involvement and increasing the contact phase. individuals with balance deficits.

During the use of the elliptical, the trunk, hip and knee maintain a greater degree of flexion, indicating greater muscle activation of the glutes and vastus lateralis, compared to walking on the ground.

In addition to the elliptical, the static bicycle, used in routine motor rehabilitation, can also be a means of training and muscle recruitment. There is movement of the knees during pedaling, the extension being the most impactful, since knee flexion is passive, as there is no greater activation of the flexors.

The pedaling variation is composed of two phases, the ascending, when the pedals move from the bottom to the top, and the descent, where the pedal displacement occurs from the top to the bottom, with greater power.

Cycling exercise can be used for muscle activation and strengthening, also performed rhythmically and alternately between the pedals. In the descending phase, there is activation of the muscles: gluteus maximus, gluteus medius, vastus intermedius, vastus lateralis, vastus medialis, rectus femoris, gastrocnemius and soleus, with hip and knee extension. In the so-called ascending phase, the ilipsoas, hamstrings and tibialis anterior muscles are activated with consequent flexion of the hip and knee.

Electromyography is a representation of the motor control of the muscular system through the placement of electrodes in the motor units and capture of electrical activity. The electromyographic analysis is used not only to verify muscle activity, but also to determine the periods of coactivation of agonist and antagonist muscles, and can assess activity for function, contraction and learning.

The electromyography signal originates from the electrical activity of the endplate. Thus, the electromyographic signal is generated by the union of the activation potentials of the motor units that are recruited concomitantly, resulting in the interference tracing.

Electromyographic biofeedback is an electronic instrument that provides information (feedback) to an individual about a physiological function or response.

ELIGIBILITY:
Inclusion Criteria:

• clinical diagnosis of spinal cord injury for at least 6 months

Exclusion Criteria:

* hip fracture
* lower limb or with pressure ulcers
* unstable angina or other decompensated heart disease
* chronic obstructive pulmonary disease,
* neurological diseases like Parkinson's,
* stroke
* Symptomatic drop in blood pressure when upright

Ages: 17 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Clinical diagnosis of spinal cord injury for at least 6 months, aged between 17 and 60 years, spastic or flaccid, of both sexes.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
comparison of muscle activation | 2 years
  difference in mean entre a atividade muscular eletromiográfica do músculo reto femoral durante 2 modalidades de exercício (andador fixo e esteira a 1 km/h, onde a diferença na média foi de 4,72 e o desvio padrão de 1,13) com poder de efeito de 90% e nível de significância de 0,05,

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Priscila Paula Dos Santos, Canoas, Rio Grande do Sul
  - Universidade Federal de Ciências da Saúde de Porto Alegre, Porto Alegre, Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: Undecided